CLINICAL TRIAL: NCT03670693
Title: Non-invasive Approaches to Identify the Cause of Fatigue in Inflammatory Bowel Disease Patients
Acronym: IBD Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17083
Record Dates: First submitted 2018-05-10; First posted 2018-09-13 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Muscle Strength; Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fatigued Crohn's Disease (Experimental): Crohns disease patients in remission(Harvey Bradshaw index <4 and CRP<5mg/dl and faecal calprotectin <50ug/g) suffering from fatigue (General fatigue and physical fatigue score on the Multiple Fatigue Inventory-20 >14, and a score of >4 in the Fatigue questionnaire.)
  Interventions: Diagnostic Test: Muscle strength and fatigue assessment; Diagnostic Test: Dual-energy X-ray absorptiometry (DEXA scan); Diagnostic Test: Supine cardiorespiratory fitness assessment; Diagnostic Test: fMRI Exercise assessment; Diagnostic Test: Muscle deconditioning assessment
- Non-Fatigued Crohn's Disease (Experimental): Crohns disease patients in remission(Harvey Bradshaw index <4 and CRP<5mg/dl and faecal calprotectin <50ug/g) without fatigue (General fatigue and physical fatigue score on the Multiple Fatigue Inventory-20 <14, and a score of <4 in the Fatigue questionnaire.)
  Interventions: Diagnostic Test: Muscle strength and fatigue assessment; Diagnostic Test: Dual-energy X-ray absorptiometry (DEXA scan); Diagnostic Test: Supine cardiorespiratory fitness assessment; Diagnostic Test: fMRI Exercise assessment; Diagnostic Test: Muscle deconditioning assessment
- Healthy Volunteers (Experimental): Age,gender,muscle mass, and physical activity-matched healthy controls.
  Interventions: Diagnostic Test: Muscle strength and fatigue assessment; Diagnostic Test: Dual-energy X-ray absorptiometry (DEXA scan); Diagnostic Test: Supine cardiorespiratory fitness assessment; Diagnostic Test: fMRI Exercise assessment; Diagnostic Test: Muscle deconditioning assessment

INTERVENTIONS:
Diagnostic Test: Muscle strength and fatigue assessment — Measurement of maximum voluntary isometric contraction of the quadricep muscle on a cybex isokinetic dynomometer. This will be followed by a fatigue assessment where the torque decrement over 20 isokinetic knee extensions at a fixed angular velocity will be quantified to assess muscle fatigue
Diagnostic Test: Dual-energy X-ray absorptiometry (DEXA scan) — Body composition will be assessed via DEXA scan (Lunar Prodigy, GE Medical Systems, Bucks, UK)
Diagnostic Test: Supine cardiorespiratory fitness assessment — VO2 peak will be quantified during completion of a continuous, incremental exercise test performed in the supine position on an MR adapted stepper machine (Ergospect, Innsbruck Austria)
Diagnostic Test: fMRI Exercise assessment — Measurement of cardiac output and, cerebral and regional perfusion using Blood-Oxygen-level-dependent (BOLD) measures and arterial spin-labelling (ASL)-MRI as well as fractional oxygen extraction using TRUST-MRI during supine exercise of the quadriceps with the MR compatible cardiostepper (Ergospect, Innsbruck, Austria) at 50% of relative VO2 peak as measured during the supine cardiorespiratory fitness assessment.
Diagnostic Test: Muscle deconditioning assessment — Limb blood flow will be occluded with a cuff, whilst participants perform repeated plantar flexion exercise in a MRI scanner. This will drive PCr, (the available reserve of ATP) to zero. Once the cuff is removed, they will undergo non-invasive and well-established in vivo 31P magnetic resonance (31P MRS) measurements on the gastrocnemius to determine PCr re-synthesis rate during resting recovery.

SUMMARY:
Crohn's disease (CD) presents with severe symptoms, but fatigue is a very predominant symptom that negatively impacts upon quality of life. Fatigue affects ~40% of patients when well and 80% of patients when the disease is active. It is the second commonest symptom that an IBD patient gets throughout their life-time. The IBD priority-setting partnership between the James Lind Alliance and the British Society of Gastroenterology has recently identified fatigue as an area of unmet clinical need and a priority research field, in which diagnosis and therapeutic intervention are lacking.

Based on other diseases that present with fatigue, the cause of fatigue may be divided into peripheral fatigue, mainly driven by anomalies in muscle mass and function and central fatigue, mainly driven through decreased blood supply to the brain during exercise probably due to decreased heart and lung fitness.

Research in IBD fatigue until now has been patchy with no convincing evidence that any treatment helps. There has been no research aimed at studying whole body function. It is imperative to have a better understanding of the alterations in muscle, brain, heart and lung function seen in these patients before specific treatments are researched.

In this study, the investigators aim to recruit 32 CD patients, half with fatigue and half without. Subjects with active disease or with other known reasons of fatigue will be excluded. Findings in this group will be compared to 16 other healthy control volunteers of a similar age, gender and Body Mass Index. The study aims to recruit all participants over 36 months, and will target people aged from 16 to 60 years of age.

Once recruited, the participants will be asked to provide their consent to take-part in 3 experiments on two separate days. These experiments have been designed to carefully consider potential fatigue burden, experimental practicality, and participant availability.

Objective 1: The investigators aim to measure muscle fitness and strength by asking subjects to exercise using a stepper, whilst body mass and composition will be measured using an X-ray. This session will take 2 hours and be undertaken on one day.

Objective 2: Peripheral fatigue: The investigators aim to non-invasively measure the recovery of muscle physiology after exercise by using magnetic resonance imaging after 5 min of exercise undertaken with a limb cuff. This will take ~1 hour.

Objective 3: Central fatigue: while in the scanner and performing exercise, the investigators aim to non-invasively measure heart and brain blood flow before and after a few minutes of exercise using magnetic resonance imaging. This will take 2 hours.

Experimental work for Objectives 2 and 3 will be undertaken on the same day. There will be ample time for recovery in between and during the different studies. There will be no further commitment from the participants required after these 2 study visits.

IBD fatigue has never been studied in such detail. This unique work will allow identification of fatigue mechanisms, which can then be targeted with exercise, nutritional, or medical treatments.

DETAILED DESCRIPTION:
Background information Inflammatory bowel disease (IBD) fatigue is, with diarrhoea, the most common medical symptom in patients with active Crohn's disease (CD) and the second commonest complaint after arthralgia in CD patients in remission. The IBD priority-setting partnership between the James Lind Alliance and the British Society of Gastroenterology has highlighted that IBD fatigue is a top 10 UK research priority.

The prevalence of fatigue ranges from 41-48% when in remission, increasing up to 86% when the disease is active. Chronic fatigue is associated with an impaired health-related quality of life in IBD and a reduced physical activity, which in paediatric cohorts plays a major role in normal growth development. In the absence of reversible clinical causes such as anaemia, inflammatory burden or nutrient deficiency, it is as yet unclear what causes fatigue in these patients. Present approaches are limited in offering clues to potential therapeutic approaches or accurate clinical evaluation for CD patients. This is likely due to a lack of a multicomponent approach and poor methodological sensitivity and reliability when assessing fatigue. A multidimensional concept of physical, cognitive and affective components have been suggested for IBD fatigue. Yet, it remains unclear how to treat IBD fatigue. Exercise therapy, psychosocial interventions and solution-focused therapy, are all suggested as treatment options but none have been shown to be convincingly effective.

Fatigue arises from peripheral and central processes, which are both equally important. While peripheral fatigue is ascribed to muscle aetiology, central fatigue is a progressive exercise-induced reduction in voluntary activation to the muscle due to failure of the central nervous system (CNS). Present approaches have been limited in failing to adequately quantify peripheral fatigue at a muscle level and central fatigue at the level of the CNS.

Peripheral fatigue: the need of muscle activity

Physical fatigue is linked to reduced muscle mass and quality (sarcopenia) and consequently reduced muscle function. Drivers of muscle mass loss include physical inactivity and anabolic resistance, which to a large extent blunt the stimulatory effect of protein nutrition on muscle protein synthesis. In keeping with this, patients with active CD show a significant decrease in expression of hypertrophy skeletal muscle signalling pathways, but no changes in the expression of atrophy signals.

Poor muscle quality is an important driver of metabolic dysfunction that is often overlooked as a driver of peripheral fatigue. In preliminary unpublished data, the investigators have shown for the first time that skeletal muscle of patients with active CD exhibits blunted glucose uptake in response to glucose feeding, suggesting diminished muscle metabolic quality in CD patients.

In fatigued IBD subjects, medium-to-large effect sizes for impaired aerobic fitness (VO2max), muscle strength and physical activity are seen in subjects with fatigue when compared to subjects with no reported history of fatigue and the normal population. Physical inactivity in quiescent CD disease could be an explanation underpinning these observations, pointing to inactivity secondary to disease burden being the aetiology of fatigue in CD, much as in chronic obstructive pulmonary disease (COPD). Physical inactivity has already been shown in CD in both paediatric and adult cohorts and has been significantly correlated to disease activity but is still prevalent in remission. Although this might imply circularity in the aetiology of fatigue in the context of physical inactivity, it is unlikely that these two factors have a simple direct cause and effect relationship. Indeed, when habitual physical activity is matched between volunteers, skeletal muscle fatigue is still most prevalent in CD, and predominantly in those subjects who complain of fatigue. Collectively, these data are indicative that both reduced cardio-respiratory fitness and peripheral muscle deconditioning (possibly linked to reduced muscle mitochondrial density) are contributing to early fatigue development in IBD patients who report symptoms of fatigue.

Central fatigue: the need of cardio-respiratory regulation

Skeletal muscle, the cardio-respiratory system and the CNS are interlinked. In preliminary data, it has been shown for the first time that it is possible to assess change of brain perfusion (or cerebral blood flow; CBF), an indirect measurement of haemodynamic measurement of brain neuronal activity, using functional MRI techniques, in relation to decreased cardiovascular fitness with age. These data have demonstrated that CBF measured directly using arterial spin labelling (ASL) or indirectly using blood-oxygen-level-dependent (BOLD) was reduced in older people with reduced cardiorespiratory fitness, and who are likely more fatigable than young volunteers. This suggests that the coupling between CBF and brain activity can be modulated by cardiac output, and thus be manipulated to improve brain function linked to central fatigue in CD patients.

This highlights the potential of non-invasive functional brain MRI techniques to determine the effect of brain perfusion during exercise on central fatigue in CD patients. Furthermore, these quantitative approaches could be used to determine whether improvements in cardiovascular fitness and appropriate downstream exercise or pharmacological interventions can alter central fatigue.

1.Aims and purpose of the proposed investigation

Hypothesis: The investigators hypothesize that the aetiology of IBD fatigue lies collectively with peripheral muscle deconditioning and brain central fatigue, the latter being secondary to a reduction in cardio-respiratory fitness and/or cardiac output, such that both central and peripheral fatigue contribute to fatigue development in IBD.

Aims:

To address this hypothesis, the investigators aim to recruit a cohort of fatigued and non-fatigued CD patients in remission and age-, gender- muscle mass-, and physical activity-matched healthy volunteers. Fatigue symptoms will be defined through relevant questionnaires at screening. The investigators will subsequently objectively quantify muscle strength of the knee extensors during a maximal voluntary isometric contraction, and fatigue development in the quadriceps muscle group. The latter will be defined as the loss in muscle peak-torque development over 20 consecutive isokinetic knee-extensions. Peripheral (muscle) and central (CNS) roles in fatigue aetiology will be investigated. Peripheral muscle deconditioning will be investigated by quantifying muscle phosphocreatine (PCr) re-synthesis during recovery from exercise using 31phosphorous MRS, while the potential of central fatigue will be examined through various measures of CNS perfusion and fractional brain oxygen extraction using MRI.

Detailed plan of investigation and scientific procedures/methodology

The investigators aim to recruit 32 patients with CD in remission, with and without a history of IBD fatigue (n=16 for IBD fatigue cohort and n=16 for no IBD fatigue cohort) within 36 months. These cohorts will be compared to 16 age-, gender- muscle mass-, and physical activity-matched healthy controls (from our existing Nottingham Digestive Diseases Biomedical Research Unit and MRC/ARUK databases) to undergo the experimental protocol outlined below. The investigators will specifically match for physical activity to investigate its potential primary effect on fatigue.

Objective 1 (Day 1): To determine muscle strength, fatigue and cardiorespiratory fitness.

Following consent, CD and healthy matched controls volunteers will perform 3 maximal isometric knee extensions of the quadriceps muscle group (each separated by 30s) to determine muscle strength. Following this, volunteers will perform 20 maximal single leg knee extensions on a Cybex isokinetic dynomometer (Cybex Norm, USA) at a constant angular velocity of 90 degrees per second to determine muscle torque development. Each maximal voluntary contraction will be initiated from a position of 90 degrees knee flexion and continued through to the point of full knee extension. After each contraction, the leg will be returned passively to the start position (approximately 1.1s) from which the next contraction will be immediately initiated. The outcome measure and the gold-standard definition of fatigue in this objective will be defined as the decline in peak torque generation for each contraction over the 20 knee extensions. Maximal voluntary contractions at this velocity has previously been shown to result in recruitment of both type I and type II muscle fibres of the quadriceps muscle group. Thirty minutes later, volunteers will undergo a continuous, incremental, supine exercise test using an MR compatible step ergometer (Ergospect diagnostic pedal). Exercise will commence at a low workload, which will increase every 3 min to determine peak VO2 during supine exercise using on-line expired gas analysis (Cosmed, Rome, Italy). Carbon dioxide (CO2) production and oxygen (O2) consumption will be measured throughout the test and used to measure peak oxygen uptake and respiratory exchange ratio (RER). These data will be normalized to body composition as measured by dual-energy X-ray absorptiometry (DEXA; Lunar Prodigy, GE Medical Systems, Bucks, UK) and will provide a gold-standard measure of cardiorespiratory (or aerobic) fitness.

Objective 2 (Day 2): To determine brain perfusion and central fatigue.

Recently, in collaboration with researchers at the Sir Peter Mansfield Imaging Centre at the University of Nottingham, the investigators have developed a protocol to quantify the cortical vascular response to exercise in volunteers and its modulation in ageing and cardiorespiratory fitness. Here, the same approach will be used to assess cortical vascular response to exercise in the brain regions associated with central fatigue of CD patients.

To study this mechanism in CD patients, the investigators propose to measure cardiac output and, cerebral and regional perfusion using Blood-Oxygen-level-dependent (BOLD) measures and arterial spin-labelling (ASL)-MRI as well as fractional oxygen extraction using TRUST-MRI respectively during supine exercise of the quadriceps with the MR compatible ergometer (Ergospect diagnostic pedal) at given values of relative VO2max (as measured in Objective 1).

This multimodal approach will determine a potential uncoupling between brain perfusion and neuronal activity and the role of central hypoxemia in central fatigue of IBD patients compared to healthy controls. Furthermore, these data will be correlated to cardiorespiratory fitness, muscle strength and fatigue, and will determine the predominant role of central processes in fatigue of IBD patients. If these brain vascular measures are associated with fatigue development, then this index of neurovascular coupling could benefit from exercise training in a similar way to muscle tissue.

Objective 3 (Day 2): To determine muscle deconditioning.

To maintain energy (ATP) during exercise, skeletal muscle regulates oxidative (mitochondrial) and non-mitochondrial production of ATP. In healthy individuals, the relative contribution of non-mitochondrial ATP production to total energy production is generally dictated by the exercise intensity, which determines the magnitude of accumulation of metabolic by-products that are directly linked to muscle discomfort and fatigue. In disease states, exacerbated fatigue and muscle pain has been attributed to reduced muscle blood flow and/or reduced mitochondrial mass.

To separate these two processes in CD patients, limb blood flow will be occluded with a cuff, whilst participants perform repeated plantar flexion exercise in a MRI scanner. This will drive PCr, (the available reserve of ATP) to zero. Specifically, participants with a lower limb cuff will perform 30 contractions over a 5-minute period using a MR compatible ergometer. Once the cuff is removed, they will undergo non-invasive and well-established in vivo 31P magnetic resonance (31P MRS) measurements on the gastrocnemius to determine PCr re-synthesis rate during resting recovery. 31P MRS data will be averaged, processed and quantified using in-house methods.

Since the rate of PCr re-synthesis is directly proportional to mitochondrial mass and oxygen delivery is not limiting during exercise recovery, this will allow us to measure muscle metabolic deconditioning in vivo.

Sample size

1. Cardiorespiratory fitness: The investigators have previously shown that the VO2max of a healthy volunteer is 3.65 (0.5) L/min, whilst the VO2max of a fatigued IBD patient is 1.99 (0.44) L/min and a non-fatigued patient is 2.43 (0.75) L/min. Assuming a power of 80% and α=0.05, 6 subjects in each group are needed to show a significant difference between the healthy volunteers and the non-fatigued cohort, and 13 patients in each group are needed to show a difference between the 2 CD cohorts.
2. Muscle Fatigue: Peak muscle Torque extension 180⁰/s (Nm) is lower in fatigued IBD vs non-fatigued IBD patients (60.73 vs 73.5, SD 12.3 respectively). Assuming a power of 90% and α=0.05, 16 CD subjects in each group are needed to show a difference between fatigued and non-fatigued CD cohorts. Importantly, the rate of muscle fatigue (defined as the gradient of force decrease from repetition 2 to 30 of an exercise protocol) is significantly greater in CD than healthy volunteers (5.2 Nm/min vs 1.3 Nm/min, SD 3. In this instance, assuming a power of 90% and α=0.05, 11 subjects in each group are needed to show a difference between CD and healthy volunteers.
3. Muscle conditioning: recent studies have shown that Pcr re-synthesis rate is 27.9 ± 0.6 s in lean sedentary subjects, whilst being 36.5 ± 2.4 s in Type 2 diabetes mellitus patients (T2DM). Thus, assuming a power of 100% and α=0.05, 3 subjects in each group are needed to show a difference between healthy volunteers and potentially fatigued cohort such as T2DM patients.
4. Anabolic resistance: Furthermore, our recent work on anabolic resistance has already shown significant differences in muscle quality between CD and healthy volunteers (significant difference observed n=5 patients). Percentage forearm fatigue in the dominant arm is 26.75%±11.1 and 18.3±7.8 in CD and controls respectively. Assuming a power of 80% and α=0.05, 11 subjects are needed in each arm.
5. MRI: It is not possible to power this exact MRI study as pilot data in these IBD cohorts has not been collected. However, the investigators have previously shown that brain perfusion in the young increases by 18±6% for 30% VO2max during a cardiorespiratory fitness test. Whilst in the elderly, it increases by only 3±4 %. Assuming a power of 100% and α=0.05, 10 subjects in each group are needed to show a significant difference between healthy volunteers (young) and a potentially fatigued cohort (elderly). Further, for fMRI BOLD analysis it is generally considered that a minimum of 12 subjects is needed in each cohort, with improved sensitivity of MR scanners (and thus higher temporal signal-to-noise ratio (SNR) now allowing improved individual subject analyses.

For the above reasons, the investigators feel that 16 subjects in each group (fatigued CD, non-fatigued CD and healthy volunteers) will suffice to show a difference in our chosen objective endpoints.

Data analysis Fatigue will be measured as the decline in peak torque development over 20 isokinetic knee extensions as described above. PCr re-synthesis rate and fractional brain oxygen extraction will be the primary endpoints in objectives 2 and 3.

31P MRS data will be analysis using standard NMR software (jMRUI Software for the clinical and biomedical MRS). Precisely, all spectra from the time series will be apodized (15-20 Hz Lorentzian shape). From these spectra, the signal intensities of 5 peaks will be determined after lineshaping. The pH will be determined prior to and at the end of the exercise protocol by measuring the frequency shift between the PCr and Pi, whilst in-house written code in MATLAB (MathWorks Inc., Matrix House, Cambridge, UK) will be used for further calculations of the PCr recovery rate. In this case, peak area intensities of the PCr peak from jMRUI will be used as input in the script to fit the data time courses using a mono-exponential function: PCr (t) = PCr (t0) + C (1 - e-t/τ); with PCr being the intensity level of the PCr peak, C a constant, τ [s] the rate constant for PCr recovery, and t [s] time, starting at the end of the exercise protocol (t0). The Reproducibility of 31P MRS measures of muscle energetics has been recently evaluated in trained human and show that coefficient of variation during exercise (27%) and at rest (8%) was relatively low, and difference were detectable with 15 volunteers. This confirms that 31P MRS approach provides reproducible and experimentally useful measures of PCr re-synthesis rate in human skeletal muscle.

BOLD MRI data will be analysed using standard neuroimaging packages (Statistical Parametric Mapping (SPM); Wellcome Department of Imaging Neuroscience and FMRIB Software Library software. Images will be motion-corrected, normalized to a standard Montreal Neurological Institute template to facilitate inter-participants averaging. For all data acquisitions, the investigators will record the vectocardiogram (VCG) and respiratory motion to allow data to be corrected for physiological noise. Contrast vectors will be formed to identify the CNS response to the exercise stimulus. The investigators will form statistical maps of those brain regions which show a decrease/increase in BOLD signal following the exercise intervention. These statistic maps will be used in contrasts by intervention and between participant groups. Results will be pooled in a second level, random effects group analysis (RFX) and active brain areas displayed at a false discovery rate corrected probability P < 0.05, k > 5. These analyses have been previously carried out and published by our group. ASL data will be motion corrected and modelled to quantify perfusion in ml/100g/min, and global and regional perfusion measures compared before and during the exercise intervention. TRUST data will be used to compute fractional oxygen extraction before and during exercise intervention. Data will be presented as mean +/- standard error of the mean (SEM). Binary comparisons will be carried out by t-tests while multiple comparisons will be carried out with an analysis of variance with a post-hoc Bonferroni correction in between the 3 groups. The effects of cytokines, vitamin D and disease duration will be investigated through a correlation co-efficient and post-hoc multivariate analysis.

The investigators will stratify subjects based on the quantitative outcome measures: PCr re-synthesis rate, cardiorespiratory fitness as measured through VO2max, decline in muscle output and change in regional perfusion and fractional brain oxygen extraction irrespective of their fatigue status. This will aid our understanding regarding which alterations in physiology and metabolism are best associated with specific fatigue symptoms. Doing this will allow objective quantification of a subjective cut-off for the IBD Fatigue scale, thereby better defining fatigue.

ELIGIBILITY:
Inclusion Criteria:

Non-Fatigued CD Patients:

* Harvey Bradshaw index <4
* CRP<5mg/dl or
* Faecal calprotectin <50ug/g or,
* As evidenced by recent endoscopy or cross-sectional imaging,
* General fatigue and physical fatigue score on the Multiple Fatigue Inventory-20 <13
* Score of <3 in the Fatigue questionnaire.

Fatigued CD Patients:

* Harvey Bradshaw index <4 and,
* CRP<5mg/dl or,
* Faecal calprotectin <50ug/g or,
* As evidenced by recent endoscopy or cross-sectional imagining and,
* General fatigue and physical fatigue score on the Multiple Fatigue Inventory-20 >14
* Score of >4 in the Fatigue questionnaire.

Inclusion criteria (Healthy volunteer participants)

* 26 Healthy Volunteers 16-75 years old matched for:
* Gender
* Muscle mass
* Physical activity
* General fatigue and physical fatigue score on the Multiple Fatigue Inventory-20 <7.

All participants should have a good command of both verbal and written English and be able to give informed consent.

Exclusion Criteria:

Exclusion criteria (CD and Healthy volunteer participants)

Potential participants with any of the following criteria will be excluded:

* >8 on the Hospital Anxiety and Depression score
* Haematological or biochemical abnormalities (e.g. anaemia (haemoglobin <13g/dl in a male and 12g/dl in a female)
* Renal failure
* Hypokalaemia
* Pregnancy or childbearing in the last 6 months
* Vitamin B complex deficiencies)
* Active or previous prescriptions of corticosteroids in the last 12 weeks
* Overt muscle wasting (defined as 2 standard deviations outside the age-related norm as measured by DEXA)
* Fatigue starting after the onset of thiopurine therapy
* Present arthritis or arthralgia
* Surgical intervention in the last 12 weeks
* Other aetiologies of chronic liver disease, specifically alcohol or drug induced liver disease, autoimmune or viral hepatitis, cholestatic or metabolic/genetic liver disease by specific clinical, biochemical, radiographic and /or histological criteria.
* Significant cardiovascular or respiratory disease
* Thyroid disease
* Current Infection
* Neurological or cognitive impairment
* Significant physical disability
* Pregnancy or breastfeeding. Participants will be informed before the DEXA scan that pregnancy is an exclusion and standard NHS procedures will be followed- pregnancy tests will be available in the female toilets of the Physiology Unit for self-testing)
* Any other conditions in addition to the above that the investigators consider may affect study measurements or safety
* Inability to understand verbal and/or written explanation of the study requirements
* >5mSv ionizing radiation exposure in the past 12 months

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Central fatigue - Cerebral perfusion | 2 hours (All central fatigue measures quantified during a single 2-hour fMRI scan)
  Cerebral perfusion will be used as a surrogate measure of central fatigue: Arterial spin labelling (ASL) data will be motion corrected and modelled to quantify brain perfusion in ml/100g/min. Both global and regional perfusion will be measured pre , during and post exercise.
Central fatigue - Oxygen extraction | 2 hours (All central fatigue measures quantified during a single 2-hour fMRI scan)
  T2 relaxation under spin tagging (TRUST) data will be used to compute fractional oxygen extraction. Data will be expressed as a percentage of cerebral blood flow and quantified pre, during and post exercise.
Central fatigue - Cardiac Output | 2 hours (All central fatigue measures quantified during a single 2-hour fMRI scan)
  Phase contrast MRI (PC-MRI) will be used to quantify realtime cardiac output. This will be quantified in the pre, during and post exercise period via quantification of heart rate and stroke volume using Phillips intellispace software. Data will be presented in L/min.
Peripheral fatigue - PCr resynthesis rate | 1 hour Magnetic Resonance Spectroscopy (MRS) scan
  Quantification of phosphocreatine (PCr) re-synthesis rate following depletion via repeated plantar flexion exercise under blood flow occluded conditions. Since the rate of phosphocreatine re-synthesis is directly proportional to mitochondrial mass and oxygen delivery is not limiting during exercise recovery, this will allow measurement of muscle metabolic deconditioning in vivo. The rate of muscle PCr resynthesis will be expressed in (mmol.kg) and plotted as a function of time. The speed of PCr recovery rate will be compared across groups and provide a gold standard measurement of muscle deconditioning and reveal any peripheral contributions to premature fatigue development.

SECONDARY OUTCOMES:
Cardiorespiratory fitness | 20 minutes
  VO2 peak obtained during an incremental supine exercise test performed on an MR compatible stepper. VO2 peak will be expressed in ml/min/kg, with a higher value reflecting an individuals ability to utilise a higher volume of oxygen during exercise.
Muscle strength | 10 minutes
  Maximum voluntary contraction performed on an isokinetic dynomometer. Torque values will be recorded in Newton-meters (NM).
Muscle fatigue | 10 minutes
  Rate of torque decrement (Newton-meters) during 20 knee extension repetitions performed on an isokinetic dynamometer at a constant angular velocity of 90 degrees per second.
General fatigue - MFI 20 | 30 minutes
  The Multiple Fatigue Inventory- 20 consists of 20 questions quantifying 20 sub-sections of fatigue. Questions 1,5,12 and 16 assess general fatigue. A higher score reflects a higher degree of fatigue. Patients scoring >14 on the general fatigue questions will be grouped into the "fatigued group" whilst patients scoring <14 will be grouped into the "non-fatigued" group. We will actively exclude any healthy volunteer participants (controls) who score >14 on the generl fatigue section of the MFI-20.
Body composition | 15 minutes
  Regional fat quantified in grams (g) via DEXA scan.
Body Composition | 15 minutes
  Lean masses quantified in grams (g) via DEXA scan.
Physical Fatigue - MFI 20 | 30 minutes
  The Multiple Fatigue Inventory- 20 consists of 20 questions quantifying 20 sub-sections of fatigue. Questions 2,8,14 and 20 assess physical fatigue. A higher score reflects a higher degree of fatigue. Patients scoring >14 on the physical fatigue questions will be grouped into the "fatigued group" whilst patients scoring <14 will be grouped into the "non-fatigued" group. We will actively exclude any healthy volunteer participants (controls) who score >14 on the physical fatigue section of the MFI-20.
Anxiety and depression - Hospital Anxiety & Depression scale (HADS) | 15 minutes
  Scores obtained from completion of the Hospital Anxiety and Depression questionnaire. This compromises separate sections of questions related to the assessment of depression and anxiety, yielding a final score for each. A higher anxiety score reflects a higher level of anxiety, whilst a lower depression score reflects more severe depression. Regarding both Anxiety & Depression scales: A score of 8-10 indicates Mild, 11-14 Moderate and 15-21 severe. We will actively exclude participants scoring >8 on either anxiety, depression, or both.
Quality of life (CUCQ-32) | 15 minutes
  Scores obtained from completion of the CUCQ-32 questionnaire can range from 0-272, where a higher score reflects a worse quality of life. There are no pre-existing, published cut off scores for this questionnaire. Mean scores will be compared across the three experimental groups to identify any differences in self-reported quality of life.
Physical activity level | 7 days
  Obtained from pedometer worn for 7 day period during the study.
Cognition | 30 minutes
  Obtained from Cognitive Assessment: Montreal Cognitive Assessment (MoCA) performed at screening. The maximum score is 30 marks, with >26 considered as normal.
Inflammatory markers | 15 minutes
  Concentrations of IL-1, IL-6, and TNFα obtained from blood sampling during screening.
Serum Vitamin D concentrations | 15 minutes
  Obtained from blood sampling during screening

CONTACTS AND LOCATIONS:
Overall Officials: Gordon W Moran, MD, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham Biomedical Research Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh S, Blanchard A, Walker JR, Graff LA, Miller N, Bernstein CN. Common symptoms and stressors among individuals with inflammatory bowel diseases. Clin Gastroenterol Hepatol. 2011 Sep;9(9):769-75. doi: 10.1016/j.cgh.2011.05.016. Epub 2011 May 20. PMID 21645640
- [Background] van Langenberg DR, Gibson PR. Systematic review: fatigue in inflammatory bowel disease. Aliment Pharmacol Ther. 2010 Jul;32(2):131-43. doi: 10.1111/j.1365-2036.2010.04347.x. Epub 2010 May 6. PMID 20456309
- [Background] Jelsness-Jorgensen LP, Bernklev T, Henriksen M, Torp R, Moum BA. Chronic fatigue is associated with impaired health-related quality of life in inflammatory bowel disease. Aliment Pharmacol Ther. 2011 Jan;33(1):106-14. doi: 10.1111/j.1365-2036.2010.04498.x. Epub 2010 Oct 25. PMID 21083587
- [Background] Tomporowski PD, Lambourne K, Okumura MS. Physical activity interventions and children's mental function: an introduction and overview. Prev Med. 2011 Jun;52 Suppl 1(Suppl 1):S3-9. doi: 10.1016/j.ypmed.2011.01.028. Epub 2011 Mar 21. PMID 21420981
- [Background] Czuber-Dochan W, Norton C, Bassett P, Berliner S, Bredin F, Darvell M, Forbes A, Gay M, Nathan I, Ream E, Terry H. Development and psychometric testing of inflammatory bowel disease fatigue (IBD-F) patient self-assessment scale. J Crohns Colitis. 2014 Nov;8(11):1398-406. doi: 10.1016/j.crohns.2014.04.013. Epub 2014 May 22. PMID 24856864
- [Background] Artom M, Czuber-Dochan W, Sturt J, Norton C. Targets for Health Interventions for Inflammatory Bowel Disease-fatigue. J Crohns Colitis. 2016 Jul;10(7):860-9. doi: 10.1093/ecco-jcc/jjw029. Epub 2016 Jan 22. PMID 26802088
- [Background] Vogelaar L, van't Spijker A, Timman R, van Tilburg AJ, Bac D, Vogelaar T, Kuipers EJ, van Busschbach JJ, van der Woude CJ. Fatigue management in patients with IBD: a randomised controlled trial. Gut. 2014 Jun;63(6):911-8. doi: 10.1136/gutjnl-2013-305191. Epub 2013 Jul 24. PMID 23884638
- [Background] Gandevia SC. Spinal and supraspinal factors in human muscle fatigue. Physiol Rev. 2001 Oct;81(4):1725-89. doi: 10.1152/physrev.2001.81.4.1725. PMID 11581501
- [Background] Schneider SM, Al-Jaouni R, Filippi J, Wiroth JB, Zeanandin G, Arab K, Hebuterne X. Sarcopenia is prevalent in patients with Crohn's disease in clinical remission. Inflamm Bowel Dis. 2008 Nov;14(11):1562-8. doi: 10.1002/ibd.20504. PMID 18478564
- [Background] Wiroth JB, Filippi J, Schneider SM, Al-Jaouni R, Horvais N, Gavarry O, Bermon S, Hebuterne X. Muscle performance in patients with Crohn's disease in clinical remission. Inflamm Bowel Dis. 2005 Mar;11(3):296-303. doi: 10.1097/01.mib.0000160810.76729.9c. PMID 15735436
- [Background] Vogelaar L, van den Berg-Emons R, Bussmann H, Rozenberg R, Timman R, van der Woude CJ. Physical fitness and physical activity in fatigued and non-fatigued inflammatory bowel disease patients. Scand J Gastroenterol. 2015;50(11):1357-67. doi: 10.3109/00365521.2015.1046135. Epub 2015 May 13. PMID 25966749
- [Background] Marimuthu K, Murton AJ, Greenhaff PL. Mechanisms regulating muscle mass during disuse atrophy and rehabilitation in humans. J Appl Physiol (1985). 2011 Feb;110(2):555-60. doi: 10.1152/japplphysiol.00962.2010. Epub 2010 Oct 28. PMID 21030670
- [Background] van Langenberg DR, Della Gatta P, Warmington SA, Kidgell DJ, Gibson PR, Russell AP. Objectively measured muscle fatigue in Crohn's disease: correlation with self-reported fatigue and associated factors for clinical application. J Crohns Colitis. 2014 Feb;8(2):137-46. doi: 10.1016/j.crohns.2013.07.006. Epub 2013 Aug 12. PMID 23938210
- [Background] Murton AJ, Marimuthu K, Mallinson JE, Selby AL, Smith K, Rennie MJ, Greenhaff PL. Obesity Appears to Be Associated With Altered Muscle Protein Synthetic and Breakdown Responses to Increased Nutrient Delivery in Older Men, but Not Reduced Muscle Mass or Contractile Function. Diabetes. 2015 Sep;64(9):3160-71. doi: 10.2337/db15-0021. Epub 2015 May 26. PMID 26015550
- [Background] Baghai-Ravary R, Quint JK, Goldring JJ, Hurst JR, Donaldson GC, Wedzicha JA. Determinants and impact of fatigue in patients with chronic obstructive pulmonary disease. Respir Med. 2009 Feb;103(2):216-23. doi: 10.1016/j.rmed.2008.09.022. Epub 2008 Nov 22. PMID 19027278
- [Background] Werkstetter KJ, Ullrich J, Schatz SB, Prell C, Koletzko B, Koletzko S. Lean body mass, physical activity and quality of life in paediatric patients with inflammatory bowel disease and in healthy controls. J Crohns Colitis. 2012 Jul;6(6):665-73. doi: 10.1016/j.crohns.2011.11.017. Epub 2012 Jan 9. PMID 22398103
- [Background] van Langenberg DR, Papandony MC, Gibson PR. Sleep and physical activity measured by accelerometry in Crohn's disease. Aliment Pharmacol Ther. 2015 May;41(10):991-1004. doi: 10.1111/apt.13160. Epub 2015 Mar 17. PMID 25783784
- [Background] Wall BT, Stephens FB, Constantin-Teodosiu D, Marimuthu K, Macdonald IA, Greenhaff PL. Chronic oral ingestion of L-carnitine and carbohydrate increases muscle carnitine content and alters muscle fuel metabolism during exercise in humans. J Physiol. 2011 Feb 15;589(Pt 4):963-73. doi: 10.1113/jphysiol.2010.201343. Epub 2011 Jan 4. PMID 21224234
- [Background] Stephens FB, Wall BT, Marimuthu K, Shannon CE, Constantin-Teodosiu D, Macdonald IA, Greenhaff PL. Skeletal muscle carnitine loading increases energy expenditure, modulates fuel metabolism gene networks and prevents body fat accumulation in humans. J Physiol. 2013 Sep 15;591(18):4655-66. doi: 10.1113/jphysiol.2013.255364. Epub 2013 Jul 1. PMID 23818692
- [Background] Greenhaff PL, Campbell-O'Sullivan SP, Constantin-Teodosiu D, Poucher SM, Roberts PA, Timmons JA. Metabolic inertia in contracting skeletal muscle: a novel approach for pharmacological intervention in peripheral vascular disease. Br J Clin Pharmacol. 2004 Mar;57(3):237-43. doi: 10.1046/j.1365-2125.2003.01989.x. PMID 14998419
- [Background] Lindeboom L, Nabuurs CI, Hoeks J, Brouwers B, Phielix E, Kooi ME, Hesselink MK, Wildberger JE, Stevens RD, Koves T, Muoio DM, Schrauwen P, Schrauwen-Hinderling VB. Long-echo time MR spectroscopy for skeletal muscle acetylcarnitine detection. J Clin Invest. 2014 Nov;124(11):4915-25. doi: 10.1172/JCI74830. Epub 2014 Oct 1. PMID 25271624
- [Background] Desmond JE, Glover GH. Estimating sample size in functional MRI (fMRI) neuroimaging studies: statistical power analyses. J Neurosci Methods. 2002 Aug 30;118(2):115-28. doi: 10.1016/s0165-0270(02)00121-8. PMID 12204303
- [Background] Edwards LM, Tyler DJ, Kemp GJ, Dwyer RM, Johnson A, Holloway CJ, Nevill AM, Clarke K. The reproducibility of 31-phosphorus MRS measures of muscle energetics at 3 Tesla in trained men. PLoS One. 2012;7(6):e37237. doi: 10.1371/journal.pone.0037237. Epub 2012 Jun 11. PMID 22701564
- [Background] Eldeghaidy S, Marciani L, McGlone F, Hollowood T, Hort J, Head K, Taylor AJ, Busch J, Spiller RC, Gowland PA, Francis ST. The cortical response to the oral perception of fat emulsions and the effect of taster status. J Neurophysiol. 2011 May;105(5):2572-81. doi: 10.1152/jn.00927.2010. Epub 2011 Mar 9. PMID 21389303
- [Background] Jenkinson M, Beckmann CF, Behrens TE, Woolrich MW, Smith SM. FSL. Neuroimage. 2012 Aug 15;62(2):782-90. doi: 10.1016/j.neuroimage.2011.09.015. Epub 2011 Sep 16. PMID 21979382
- [Background] Glover GH, Li TQ, Ress D. Image-based method for retrospective correction of physiological motion effects in fMRI: RETROICOR. Magn Reson Med. 2000 Jul;44(1):162-7. doi: 10.1002/1522-2594(200007)44:13.0.co;2-e. PMID 10893535
- [Background] Jones RB, McKie S, Astbury N, Little TJ, Tivey S, Lassman DJ, McLaughlin J, Luckman S, Williams SR, Dockray GJ, Thompson DG. Functional neuroimaging demonstrates that ghrelin inhibits the central nervous system response to ingested lipid. Gut. 2012 Nov;61(11):1543-51. doi: 10.1136/gutjnl-2011-301323. Epub 2012 Feb 7. PMID 22315469
- [Background] Lassman DJ, McKie S, Gregory LJ, Lal S, D'Amato M, Steele I, Varro A, Dockray GJ, Williams SC, Thompson DG. Defining the role of cholecystokinin in the lipid-induced human brain activation matrix. Gastroenterology. 2010 Apr;138(4):1514-24. doi: 10.1053/j.gastro.2009.12.060. Epub 2010 Jan 18. PMID 20080096